CLINICAL TRIAL: NCT01600196
Title: Surgical Resection Versus Best Supportive Care for Resectable Hepatocellular Carcinoma Invading the First Branch of Portal Vein
Brief Title: Resection vs. Best Supportive Care for Hepatocellular Carcinoma (HCC) With Portal Venous Thrombus
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangzhou 8th People's Hospital (Other); Kaiping Central Hospital (Other); The 458 Hospital of Chinese People's Liberation Army (Unknown)
Responsible Party: Principal Investigator, Shi Ming, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC2005009
Record Dates: First submitted 2012-05-13; First posted 2012-05-16 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Hepatocellular Carcinoma With Portal Vein Tumor Thrombus
Keywords: Hepatectomy; Thrombectomy; Hepatocellular carcinoma; Portal vein tumor thrombus
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Hepatectomy; Thrombectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resection arm (Experimental): Liver resection Plus Thrombectomy
  Interventions: Procedure: Liver resection plus Thrombectomy
- Best support care arm (No Intervention): Best supportive care

INTERVENTIONS:
Procedure: Liver resection plus Thrombectomy — Liver resection plus Thrombectomy
  Other Names: Removal of all tumor tissue by surgery
  Arms: Resection arm

SUMMARY:
The purpose of this study is to evaluate the long-term efficacy and safety of surgical resection compared with best supportive care in patients with resectable hepatocellular carcinoma (HCC) with portal venous thrombus (PVTT) in the first branch of portal vein.

DETAILED DESCRIPTION:
Advances in surgical techniques have made it possible to remove all macroscopic tumors in more hepatocellular carcinoma (HCC) patients with portal venous thrombus (PVTT). However, the benefit of such surgery remains largely controversial. On one hand, many clinicians believe that surgical resection offers the only chance for long term survival. Many studies reported a median survival of 6-40 months after liver resection and thrombectomy, and some cases achieved long term survival.On the other hand, the strength of evidences arising from these studies was widely questioned because of their retrospective nature and study design. Most of them were single arm cohort study. A few studies used control groups consisted of patients with unresectable HCC and PVTT underwent transarterial chemoembolization. This led to obvious selection bias. Because patients with unresectable HCC and PVTT have a much poorer prognosis compared with resectable disease because of more widespread tumor focus and less residual liver, even if their baseline characters are comparable.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of HCC was made according to AASLD guidelines
* Main tumor ≥ 7 cm
* Imaging confirmed the presence of PVTT in the first branches but not
* Extend into the main trunk of portal vein
* Eastern Co-operative Group performance
* Resectable disease

Exclusion Criteria:

* Child-Pugh class B or C liver cirrhosis
* An American Society of Anesthesiologists (ASA) score ≥ 3
* Extrahepatic metastasis
* Patients had access to sorafenib.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2006-01; Primary Completion 2009-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Survival time | 5-years

SECONDARY OUTCOMES:
Number of Adverse Events | 30 days
  Number of adverse events, and number of patients who developed adverse event. Postoperative adverse events were graded based on the Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, MD., Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Le Treut YP, Hardwigsen J, Ananian P, Saisse J, Gregoire E, Richa H, Campan P. Resection of hepatocellular carcinoma with tumor thrombus in the major vasculature. A European case-control series. J Gastrointest Surg. 2006 Jun;10(6):855-62. doi: 10.1016/j.gassur.2005.12.011. PMID 16769542
- See also: web site of Cancer Center, Sun Yat-sen University — http://www.sysucc.org.cn